CLINICAL TRIAL: NCT02276430
Title: A Case-cohort Study to Identify Risk Factors for Cardiovascular Disease in Testicular Cancer Survivors
Brief Title: TACkLE Study - Tackling Adverse Chemotherapy-associated Late Effects
Acronym: TACkLE
Status: Active, not recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: KWF2011-5209; NL45655.042.13 (Other: ABR form)
Record Dates: First submitted 2014-07-31; First posted 2014-10-28 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Testicular Cancer
Keywords: Testicular cancer; Survivor; Cardiovascular disease; Risk factors
MeSH Terms: conditions — Testicular Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples: analysis of cardiovascular risk factors (lipid profile, glucose metabolism, hormonal status), platinum levels and several biomarkers.
  Urine samples: microalbuminuria, platinum levels. DNA: polymorphisms in candidate genes for development of cardiovascular damage, leukocyte telomere length
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: Patients who developed cardiovascular disease after testicular cancer treatment
  Interventions: Other: Vena punction
- Subcohort members: A random selection out of the total cohort of testicular cancer patients per participating hospital
  Interventions: Other: Vena punction

INTERVENTIONS:
Other: Vena punction — Once 90 ml

SUMMARY:
Testicular cancer (TC) is a rare disease, which mostly affects young men aged 15-35 years. Their life expectancy has greatly improved due to the introduction of platinum-containing chemotherapy for disseminated TC in the late 1970s. Given the good prognosis of TC nowadays, prevention or early detection of late adverse effects of TC treatment has become increasingly important. Current literature suggests that TC treatment, and specifically exposure to platinum agents, is associated with increased risk of cardiovascular morbidity and mortality. The precise role of treatment components like platinum in the pathogenesis of cardiometabolic changes and cardiovascular disease (CVD) warrants further investigation, since it is not known if CVD develops through direct platinum-induced damage of the vascular wall or by mediation through development of cardiometabolic riskfactors. The aim of this study is to identify risk factors for development for CVD after treatment for TC. A more profound insight into pathophysiologic mechanisms and identification of risk factors for CVDs is needed to facilitate development of preventive strategies and to optimize survivorship care.

DETAILED DESCRIPTION:
Design: The investigators will perform a multicenter case-cohort study. Patients treated for TC who developed cardiac disease ((either myocardial infarction, proven coronary artery disease (grade ≥2) or congestive heart failure (grade ≥2)) will be invited by their (former) treating oncologist to participate in this study (cases). Furthermore, in each hospital a random sample of 15% of the total population treated for TC will be invited (the subcohort). The investigators will collect detailed diagnostic- and treatment data on TC and on (risk factors for) CVD for all cases as well as for all subcohort members. All cases and subcohort members will be approached to complete a questionnaire and to donate a blood sample for DNA analysis, after written informed consent. Patients who were younger than 40 years at TC diagnosis and younger than 75 years at moment of study contact will be asked to participate in the cardiometabolic risk inventory sub study. For this, participants have to undergo a basic study assessment consisting of physical examination, venapuncture and handing in a morning urine sample. This assessment can be performed at the participating hospital, their general practitioner or during a home visit by a member of the investigators research team. Additional (non-invasive) cardiovascular function measurements (IMT and AGEs) are only performed in the UMCG.

ELIGIBILITY:
All participating patients have to meet the following criteria:

* Alive
* TC diagnosis between 01-01-1976 to 31-12-2007
* TC treatment center: UMCG, NKI/AVL, Erasmus MC, UMCN, LUMC
* Younger than 50 years of age at TC diagnosis
* Written informed consent

Cases have to fulfill, beside the aforementioned criteria, the following criteria:

* Diagnosed with either myocardial infarction (MI), proven coronary artery disease (CAD) (CTCAE-4 grade 2 or higher) or congestive heart failure (CHF) (CTCAE-4 grade 2 or higher).
* No medical history of CVD before diagnosis of TC

In order to be eligible to participate in the cardiometabolic risk inventory study (and to be invited to a study assessment), a subject must meet, next to the criteria mentioned in "1)", the following inclusion criteria:

* Younger than 40 years of age at TC diagnosis
* Younger than 75 years of age at moment of inclusion

Exclusion criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Mental disorder (no informed consent available)
* Presence of active malignant disease

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Testicular cancer survivors
Sampling Method: Probability Sample
Enrollment: 939 (Actual)
Dates: Start 2014-07; Primary Completion 2017-05-08 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Characteristics of disease (i.e. stage/IGCCCG prognosis group) and treatment (chemotherapy/radiotherapy) | 4 years
  To evaluate the independent and joint effects of disease- and treatment characteristics of TC patients on cardiovascular disease risk.
Cardiovascular risk factors | 4 years
  To evaluate the effect of cardiometabolic risk factors (presence of metabolic syndrome, smoking behaviour, obesity, hypertension, dyslipidemia, diabetes mellitus, family history, physical activity) on cardiovascular disease risk in TC patients.

SECONDARY OUTCOMES:
Biomarkers for endothelial activation, hemostatic activity and inflammatory activity after TC treatment and relation with CVD | 4 years
  To determine endothelial activation, hemostatic activity and inflammatory activity (represented by circulating biochemical markers) years after treatment for TC and its relationship between development of (components of) the metabolic syndrome and development of cardiovascular diseases.
Hypogonadism after TC treatment and relation with CVD | 4 years
  To evaluate the presence of hypogonadism in TC survivors and to investigate the association between hypogonadism and presence of (components of) the metabolic syndrome and development of cardiovascular disease.
DNA and telomere length analysis and association with (riskfactors for) CVD | 4 years
  To investigate the presence of candidate single nucleotide polymorphisms in genomic DNA and telomere length and its association with presence of (components of) the metabolic syndrome and development of cardiovascular disease.
Quality of life | 4 years
  To investigate the impact of cardiovascular disease on Quality of Life (QoL) in TC survivors.
Circulating platinum levels | 4 years
  In patients treated with platinum-containing chemotherapy: to evaluate circulating platinum levels in TC survivors and to investigate the relationship between circulating platinum levels and presence of (components of) the metabolic syndrome and development of cardiovascular disease.
Intima media thickness | 4 years
  Patients visiting the UMCG for the study visit: to evaluate thickness of the intima media of the carotid artery as a marker for subclinical damage in TC survivors, and to investigate the relationship between abnormal intima media thickness and presence of (components of) the metabolic syndrome and development of cardiovascular disease.
Arterial stiffness | 4 years
  Patients visiting the UMCG for the study visit: to assess the elasticity of the arterial wall of the carotid artery in TC survivors, and to investigate the relationship between abnormal arterial stiffness and presence of (components of) the metabolic syndrome and development of cardiovascular disease.
Skin auto fluorescence (SAF) as measure for Advanced Glycation End products (AGEs) | 4 years
  Patients visiting the UMCG for the study visit: to assess levels of AGEs with help of the SAF in TC survivors and to to investigate the relationship between SAF and presence of (components of) the metabolic syndrome and development of cardiovascular disease.

CONTACTS AND LOCATIONS:
Overall Officials: J. A. Gietema, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (3):
- Netherlands (3):
  - Antoni van Leeuwenhoek Hospital, Amsterdam
  - University Medical Center Groningen, Groningen
  - University Medical Center St. Radboud, Nijmegen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lubberts S, Groot HJ, de Wit R, Mulder S, Witjes JA, Kerst JM, Groenewegen G, Lefrandt JD, van Leeuwen FE, Nuver J, Schaapveld M, Gietema JA. Cardiovascular Disease in Testicular Cancer Survivors: Identification of Risk Factors and Impact on Quality of Life. J Clin Oncol. 2023 Jul 1;41(19):3512-3522. doi: 10.1200/JCO.22.01016. Epub 2023 Apr 18. PMID 37071834